CLINICAL TRIAL: NCT04647682
Title: Feasibility and Effect of Implementing Physical Activity Program Implementation During COVID-19 in Hospitalized Positive COVID-19 Older Adults
Brief Title: Physical Activity Program Implementation in Hospitalized Positive COVID-19 Older Adults
Acronym: Cov-activity
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0145
Record Dates: First submitted 2020-10-29; First posted 2020-12-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Infection
Keywords: older adults; hospital; physical activity program
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One single group study: Patients aged 75 years and over Hospitalized in a French COVID-19 geriatric unit Positive COVID-19 infection made by Real-time Polymerase Chain Reaction COVID-19 or suspected on thoracic lesions on computerized tomography.
  Interventions: Other: physical activity program

INTERVENTIONS:
Other: physical activity program — * 30 second chair test,
  * balance with joint-feet and semi-tandem stance
  * 4 meters comfortable walking test were evaluated

SUMMARY:
Our hypothesis was that physical activity program will be acceptable and may counteract physical and mental decline among older adults hospitalized in COVID-19 unit

DETAILED DESCRIPTION:
The 30 second chair test, balance with joint-feet and semi-tandem stance, and 4 meters comfortable walking test were evaluated. Depending on their score, a specific physical activity (PA) program was selected and explained. The program was printed, explained and left in the room. This intervention included 5 different PA programs.

Final evaluation (one day before leaving the unit) recording physical performance (same physical tests used for inclusion evaluation), Hospital Anxiety and depression (HAD) score, Activities Daily Living (ADL) and self-satisfaction of the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years and over
* Hospitalized in a French COVID-19 geriatric unit
* Positive COVID-19 infection made by Real-time Polymerase Chain Reaction COVID-19 or suspected on thoracic lesions on computerized tomography.

Exclusion Criteria:

* Exclusion of patients of palliative care,
* Severe dementia or Mini Mental State Examination (MMSE) [14] below 18/30
* Acute COVID-19 complication.
* Activities of Daily Living < 2/6

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Included in a French COVID-19 geriatric unit in Toulouse, hospitalized for a positive COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Change of adherence of the intervention | through study completion, an average of 15 days
  adherence of the intervention evaluated by the number of completed exercise days compared to the number of total intervention days

SECONDARY OUTCOMES:
Change of physical performances | through study completion, an average of 15 days
  Comparison between inclusion and final physical performances measured by the 30-second chair test, balance with joint-feet, semi-tandem stance, 4 meters comfortable walking test, functional abilities with the evaluation of ADL score and HAD scores.

CONTACTS AND LOCATIONS:
Overall Officials: Yves ROLLAND, MD, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (2):
  - CHU de Grenoble, Grenoble
  - University Hospital Toulouse, Toulouse
- CHU Pointe-à-Pitre Abîmes - GUADELOUPE, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andre L, Rolland Y, Gerard S, Kergoat MJ, Peyrusque E, Aubertin-Leheudre M. Feasibility and Effect of Implementing Physical Activity Program Implementation during Covid-19 in Hospitalized Positive Covid-19 Older Adults. J Nutr Health Aging. 2021;25(6):724-726. doi: 10.1007/s12603-021-1596-4. No abstract available. PMID 34179924